CLINICAL TRIAL: NCT04231292
Title: A Multicenter, Randomized, Single-blind, Active Comparator Controlled Phase 2 Clinical Study on the Effectiveness, Safety and Pharmacokinetics of Pegerythropoietin Injection (RD01) in Different Medication Schemes for the Treatment of Anemia in Chronic Renal Failure Patients With Hemodialysis
Brief Title: A Phase 2 Clinical Study of Pegerythropoietin Injection (RD01) for the Treatment of Anemia in Chronic Renal Failure Patients With Hemodialysis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shengzhen Sciprogen Bio-pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SZSBE-RD01-HD-II-01
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Patient of Anemia in Chronic Renal Failure With Hemodialysis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Experimental Group A +Group a (Experimental): Group A: 0.8μg/kg RD01, once every two weeks, Day 1~ 18th week;Group a: refers to the weekly dose at the end of the first stage , once every two weeks, 19th~46th week
  Interventions: Drug: RD01
- Experimental Group B +Group b (Experimental): Group B: 1.2μg/kg RD01, once every two weeks, Day 1~ 18th week; Group b: refers to the weekly dose at the end of the first stage , once every four weeks, 19th~46th week
  Interventions: Drug: RD01
- Experimental Group C +Group c (Experimental): Group C: 1.6μg/kg RD01, once every two weeks, Day 1~ 18th week; Group c: refers to the weekly dose at the end of the first stage , once every six weeks, 19th~46th week
  Interventions: Drug: RD01
- Experimental Group D +Group d (Experimental): Group D: 0.8μg/kg RD01, once every two weeks, Day 1~ 18th week; Group d: refers to the weekly dose at the end of the first stage , once every four weeks, 19th~46th week
  Interventions: Drug: RD01
- Experimental Group E +Group e (Active Comparator): Group E: 150IU/kg rHuEPO, once a weeks, subcutaneous administration, Day 1~ 18th week; Group e: refers to the weekly dose at the end of the first stage , once a weeks, intravenous administration, 19th~46th week
  Interventions: Drug: Recombinant Human Erythropoiesis Injection (CHO cell)
- Experimental Group F +Group f (Placebo Comparator): Group F: 8μl placebo, once every two weeks, for 6 weeks; 150 IU/kg rHuEPO, once week, subcutaneous injection, 7th ~ 18th week; Group f: refers to the weekly dose at the end of the first stage , once a weeks, subcutaneous administration, 19th~46th week
  Interventions: Drug: Recombinant Human Erythropoiesis Injection (CHO cell); Drug: placebo
- Experimental Group G (Experimental): Group G: 1.6μg/kg RD01, once every four weeks, Day 1~ 28th week;
  Interventions: Drug: RD01

INTERVENTIONS:
Drug: RD01 — RD01 is a PEGylated recombinant human erythropoietin with the same biological effects as natural erythropoietin
  Other Names: pegerythropoietin Injection
  Arms: Experimental Group A +Group a; Experimental Group B +Group b; Experimental Group C +Group c; Experimental Group D +Group d; Experimental Group G
Drug: Recombinant Human Erythropoiesis Injection (CHO cell) — rHuEPO is a recombinant human erythropoietin with the same biological effects as natural erythropoietin
  Other Names: rHuEPO
  Arms: Experimental Group E +Group e; Experimental Group F +Group f
Drug: placebo — placebo
  Arms: Experimental Group F +Group f

SUMMARY:
A multicenter randomized, single blind, active comparator controlled phase 2 study which is to evaluate the effectiveness, safety and the PK/PD characteristics of different doses, frequencies and routes of pegerythropoietin Injection (RD01) as maintenance therapy in the treatment of anemia in chronic renal failure patients with hemodialysis

DETAILED DESCRIPTION:
This trial is a multicenter randomized, single blind, active comparator controlled phase 2 study. The study is divided into two stages. The first stage lasts for 18 weeks, and is divided into fixed dose period (day 1~ 6th week ) and dose adjustment period (7th ~ 18th week). The second stage lasts for 28 weeks, and is also divided into dose adjustment period (19th ~ 38th week) and evaluation period (39th ~ 46th week).

Patients are randomly assigned to seven study groups in the first stage. Of all these seven groups, six groups are: Group A (0.8μg/kg RD01, once every two weeks, subcutaneous injection, for 18 weeks)、Group B (1.2μg/kg RD01, once every two weeks, subcutaneous injection, for 18 weeks)、Group C (1.6μg/kg RD01, once every two weeks, subcutaneous injection, for 18 weeks)、 Group D (0.8ug/kg RD01, once every two weeks, intravenous injection, for 18 weeks)、Group E ( 150 IU/kg rHuEPO, once a week, subcutaneous injection, for 18 weeks )、Group F (8μl /kg placebo, once every two weeks, for 6 weeks; then 150 IU/kg rHuEPO, once a week, subcutaneous injection, 7th ~ 18th week ).

At the beginning of the second stage, some patients in these six goups need to be be randomized again. Of which patients in Group A、B、C are randomly assigned to Group a ( RD01, once every two weeks, subcutaneous injection, 19th ~ 46th week )、Group b (RD01, once every four weeks, subcutaneous injection, 19th ~ 46th week)、Group c (RD01, once every six weeks, subcutaneous injection, 19th ~ 46th week); Patients in Group D enter directly to Group d (RD01, once every four weeks, intravenous injection, 19th ~ 46th week); Patients in Group E and F are randomly assigned to Group e (rHuEPO once a week, intravenous injection, 19th ~ 46th week ) and Group f (rHuEPO once a week, subcutaneous injection, 19th ~ 46th week). The starting dose of the second stage for individual patient in all groups refers to the weekly dose at the end of the first stage .

During the whole study period, all patients in six groups are not allowed to adjust dosage in the first 6 weeks, while in the remaining trial period dosage adjustment was allowed once every two weeks if necessary.

There is a special Group G (1.6μg/kg RD01, once every four weeks, subcutaneous injection, Day 1 ~ 28th week), all patients are allowed to adjust dosage during the whole 28 weeks.

This phase 2 study is to evaluate the effectiveness, safety and the PK/PD characteristics of different doses, frequencies and routes of pegerythropoietin Injection (RD01) as maintenance therapy in the treatment of anemia in chronic renal failure patients with hemodialysis

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic renal failure who are undergoing maintenance hemodialysis for at least 12 weeks;
* 18 ≤ age ≤ 75 years of age, male or female;
* Patients who have received short-acting EPO treatment and meets the treatment standard (hemoglobin 100 ~ 120 g / L). The mean Hb value in the screening period (at least two weeks apart ) is within the range of 100 ~ 120 g / L (both ends). The difference is less than 10g / L;
* Evaluation of iron status during the screening period, transferrin saturation (TSAT) ≥20% or serum ferritin (SF) ≥200 μg / L;
* Evaluation of dialysis adequacy during the screening period, with SpKt / V≥1.2 or URR≥65%;
* Subjects agree to use reliable contraceptives from the screening period to within 6 months after the last medication
* Sign the informed consent.

Exclusion Criteria:

* Patients who have received or plan to have a kidney transplant during the study period
* Except of renal anemia, there are other diseases that cause chronic anemia (such as sickle cell anemia, myelodysplastic syndrome, hematological malignancies, myeloma, hemolytic anemia, pure red blood cell aplastic anemia)
* Patients with acute or chronic blood loss (such as upper gastrointestinal bleeding) in the past 3 months or patients who have undergone surgery with extensive bleeding, or patients who plan to undergo surgery during the study period
* Patients with coagulation dysfunction (time to activate partial thromboplastin> 1.5 times the upper limit of normal value)
* The following circumstances (including but not limited to) during the screening, investigators evaluated that it is not suitable for enrollment:

  1. Abnormal liver function (aspartate aminotransferase or alanine aminotransferase is more than 3 times the upper limit of normal value);
  2. Patients who were positive for Hepatitis B surface antigen (HBsAg), hepatitis B core antigen (HBeAg), HIV antibody (HIV-Ab), hepatitis C virus antibody (HCV-Ab) or Treponema pallidum antibody;
* Patients with severe secondary hyperparathyroidism (iPTH> 1000 ng / L);
* Patients with severe hypertension and poor control of blood pressure (systolic blood pressure> 180 mmHg or diastolic blood pressure> 100 mmHg)
* Patients with severe thromboembolic disease
* People with severe cardio-cerebral vascular disease (excluding luminal infarction), severe or unstable coronary artery disease, heart failure (NYHA III or IV) or myocardial infarction or stroke within 3 months
* Patients with malignant tumors (excluding non-melanoma skin cancer or resected cancer in situ)
* People with a history of severe allergies (including drug allergies), allergies to erythropoietin, or allergic to any component of the test drug (such as human serum albumin)
* People with severe infection who are receiving systemic antibiotics
* Patients who have received androgen therapy or blood transfusion therapy within the last 8 weeks;
* Participated in other new drug clinical trials as a subject within 3 months or the withdrawal time was shorter than the 5 half-life of the test drug at the time of enrollment (whichever is the longest);
* Patients with a history of seizures
* Pregnant and lactating women
* Alcohol, drug or drug addicts
* Other situations that the researcher believes may affect validity judgment or are not suitable for participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy index : The change of hemoglobin concentration of experimental group from baseline to the end of 4th and 6th week | Day 1~4th week & Day 1~6th week
Primary efficacy index: The difference of hemoglobin concentration between the experimental group and the placebo group at the end of 4th and 6th week; | Day 1~4th week & Day 1~6th week
Primary efficacy index: hemoglobin concentration change from baseline to the end of first stage | Day 1~18th week
  The amount of change in hemoglobin concentration from baseline to the end of the first stage
Primary efficacy index: hemoglobin concentration change from baseline to the evaluation periods in the second stage (39th ~46th week) | Day 1~ evaluation periods (39th ~46th week)
  The amount of change in hemoglobin concentration from baseline to the evaluation periods in the second stage (39th ~46th week).

SECONDARY OUTCOMES:
Secondary efficacy index: the optimal dosage | the end of 18th week & 39th ~46th week
  The optimal dosage of the subjects at the end of the first stage and the evaluation period (39th ~46th week) in the second stage
Secondary efficacy index: maintenance rate | 39th-46th week
  the proportion of subjects whose average Hb concentration remain within the target range during the evaluation period
Secondary efficacy index : Proportion of subjects with unstable Hb during the evaluation period | 39th-46th week
Secondary efficacy index: proportion of times of Hb remains within the target range | 39th-46th week
  the proportion of times the measured Hb concentration remains within the target range during the evaluation period;
Secondary efficacy index: EPO dose conversion coefficient of RD01 | end of 18th week & 39th ~46th week
  EPO dose conversion factor for subjects at the end of the first stage and evaluation periods in the second stage
Safety indicator: adverse events | for 46 weeks
  the type, proportion and severity of adverse events
Immunogenicity indicator: incidence of anti-RD01 antibodies | for 46 weeks
  incidence of anti-RD01 antibodies
Maximum Plasma Concentration (Cmax) | for 46 weeks
  the Cmax of RD01 in patients with long-term medication.
Area Under the Curve (AUC) | for 46 weeks
  the AUC of RD01 in patients with long-term medication.

CONTACTS AND LOCATIONS:
Locations (1):
- Renal Rheumatology and Immunology department Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided